CLINICAL TRIAL: NCT01413698
Title: Cough Count Validation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Prof. Noam Gavriely MD, PhD., KarmelSonix Ltd.
Other Study IDs: KSI-IL-HHZ-CCF-01
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patient with chronic cough

SUMMARY:
People with respiratory infection, asthmatic patients and cystic fibrosis (CF) patients suffer from a multitude of pathologies of airways and are often inflicted with chronic cough.

Treatment of cough in these patients consists of many types of expectorants, cough suppressors, secretion modifiers, inhaled bronchodilators etc. In addition, chest physical therapy (PT) is often prescribed as part of the treatment regime.

The assessment of coughing is currently subjective and based on the symptoms qualitative description as expressed by the patient or parent. Quantitative and objective methods for cough assessment are not available beyond the investigative laboratory and are unique to the specific investigator.

DETAILED DESCRIPTION:
Cough is part of the defense mechanism to protect the lung from foreign particles and remove secretions from the airways . While the cough reflex is essential in protecting the lung from foreign materials and infection, its excessive or chronic presence is both bothersome and might interfere with the quality of life, sleep pattern and exercise tolerance of the patient. Such a symptom may potentially be indicative of an on-going pathological process , .

People with respiratory infection, asthmatic patients and CF patients suffer from a multitude of pathologies of airways and are often inflicted with chronic cough.

Treatment of cough in these patients consists of many types of expectorants, cough suppressors, secretion modifiers, inhaled bronchodilators etc. In addition, chest physical therapy (PT) is often prescribed as part of the treatment regime.

The assessment of coughing is currently subjective and based on the symptoms qualitative description as expressed by the patient or parent. Quantitative and objective methods for cough assessment are not available beyond the investigative laboratory and are unique to the specific investigator.

The primary objective of the study is to evaluate the efficacy and validity of novel cough counting device based on the WIM Technology.

The PulmoTrack™ technology includes the PulmoTrack™ 3010/5050 devices that are intended for the analysis, interpretation and recording of lung sounds, and the Automatic Cough Counting Application.

The recording of the lung sounds will be performed by a PulmoTrack™ 3010/5050 device. The lung sounds can subsequently be analyzed for the presence of wheezes and for the presence of cough by the Automatic Cough Counting Application (ACCA).

The technology enables accurate cough count and timing as well as wheeze detection over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-80 years.
* Patients with significant chronic cough.
* Patients in hemodynamic stability. Patient is not in respiratory distress.
* Subject or subject's parents/guardians is able to comprehend and give informed consent for participation in the study.

Exclusion Criteria:

* Contraindication to the use of the PulmoTrack™ or performing ARM (Acoustic Respiratory Monitoring).
* Hemodynamic instability and/or SOB.
* Concurrent additional major illness.
* Concurrent participation in any other study.
* Physician objection

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic cough
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Cough count | recording lasting up to 24 hours

SECONDARY OUTCOMES:
WheezeRate (the proportion of wheezing in the respiratory cycle) , respiratory rate, Inspiratory/Expiratory ratio, SPO2, symptom score (according to a questioner) | recording lasting up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Israel